CLINICAL TRIAL: NCT05732129
Title: The Efficacy and Safety of Fluzoparib Combined With Fluzoparib as Second-line Treatment in Patients With Homologous Recombination Deficiency (HRD) Metastatic Colorectal Cancer: A Single-center, Open-label, Single-arm Study .
Brief Title: The Efficacy and Safety of Fluzoparib Plus Irinotecan as Second-line Treatment in Patients With Homologous Recombination Deficiency (HRD) Metastatic Colorectal Cancer.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ye Xu, Professor, Chief of Department of Colorectal Surgery, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2207257-12
Record Dates: First submitted 2023-02-08; First posted 2023-02-16 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Homologous Recombination Deficiency Alterations Metastatic Colorectal Cancer
Keywords: Fluzoparib Plus Irinotecan; Homologous Recombination Deficiency (HRD) Alterations
MeSH Terms: conditions — Kenny-Caffey syndrome, Type 1 | interventions — fluzoparib; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fluzoparib plus Irinotecan (Experimental): Patients will receive Fluzoparib combined with Irinotecan treatment protocol, which included irinotecan asintravenous infusion at 180mg/m2 (on day 1) and Fluzoparib 150mg capsules given bid (days 1-7) every 2 weeks .
  Interventions: Drug: Fluzoparib; Drug: Irinotecan

INTERVENTIONS:
Drug: Fluzoparib — 150mg,orally, bid (days 1-7) every 2 weeks
Drug: Irinotecan — 30-90min continuous infusion 180mg/m2 Irinotecan on day 1, q2w

SUMMARY:
Preclinical data support the investigation of PARP inhibitors in other neoplasms exhibiting homologous recombination deficiency (HRD) as monotherapy as well as in combination with chemotherapy. However，in colorectal cancer (CRC), the role of HRD alterations is mostly unknown. This study aims to explore the the Efficacy and Safety of Fluzoparib combined with Irinotecan in the Second-line treatment of HRD alterations metastatic colorectal cancer.

DETAILED DESCRIPTION:
Study protocol for an open-label, single-arm, phase II study of combination of Fluzoparib and rinotecan as the second-line treatment for patients with HRD alterations metastatic colorectal cancer (mCRC). Patients will receive Fluzoparib combined with Irinotecan treatment protocol, which included irinotecan asintravenous infusion at 180mg/m2 (on day 1) and Fluzoparib 150mg capsules given bid (days 1-7) every 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years；
* Histological or cytological confirmed metastatic colorectal cancer;
* HRD alterations（inclued BRCA1/2、ATM、CDK12、PALB2、Check2、RAD51C、RAD51D etc.）；
* Intolerability toxicity occurs 8 weeks within first-line therapy;
* ECOG PS 0-1;
* Adequate hepatic, renal, heart, and hematologic functions;
* Negative serum pregnancy test at screening for women of childbearing potential;
* Informed consent was signed before the study began.

Exclusion Criteria:

* Prior treatment with PARPi drugs；
* Symptomatic brain or meningeal metastases；
* Patients have received local radiotherapy within 1 month prior to treatment;
* Patients who had active bleeding or coagulopathy before enrollment, had a tendency to bleed, or were receiving thrombolytic therapy and were considered by the investigator to be ineligible for enrollment;
* Women who are pregnant (with a positive pregnancy test before medication) or breastfeeding;
* Expected survival <3 months;
* Received other investigational drugs within 4 weeks prior to treatment;
* Patients who had active uncontrollable neurological, mental disease or mental disorder, poor compliance, unable to cooperate and describe the treatment response;
* Allergy to the study drug or any of its excipients;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate of Metastatic Colorectal Cancer,inculdthe proportion of patients with complete response or partial response | assessed up to 1 year
  using RECIST v 1.1.

SECONDARY OUTCOMES:
Progression-Free Survival of Metastatic Colorectal Cancer，includ time from enrollment to the first documented disease progression or death due to any cause, whichever occurs first | assessed up to 1 year
  Responses are according to the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by investigator
Overall survival of Metastatic Colorectal Cancer, include time from randomization to death from any cause | assessed up to 2 year
  Responses are according to the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by investigator
The Safety of Fluzoparib Plus Irinotecan as Second-line Treatment in Patients With Homologous Recombination Deficiency (HRD) Metastatic Colorectal Cancer. | assessed up to 2 year
  time from enrollment to the first documented disease progression or death due to any cause, whichever occurs first. Responses are according to the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by investigator

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Colorectal Surgery Fudan University Shanghai Caner Center, Shanghai, Shanghai Municipality, China